CLINICAL TRIAL: NCT05906355
Title: A Prospective, Cross-over, Controlled Primary Clinical Evaluation of the Precision, Security, and Operability of Wearable Filtrating Artificial Kidney Device for On-site Medical Rescue
Brief Title: Primary Clinical Evaluation of Wearable Filtrating Artificial Kidney Device for On-site Medical Rescue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jianhui Zhou, Professor, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S2022-120-01
Record Dates: First submitted 2023-01-31; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Fluid Overload
Keywords: Wearable; Artificial Kidney Device; Fluid Overload
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A（wearable filtrating artificial Kidney+traditional hemodialysis） (Experimental): Group A was isolated ultrafiltration with wearable filtrating artificial Kidney Device first, and then with traditional hemodialysis machine.
  Interventions: Device: the wearable filtrating artificial Kidney Device; Device: traditional hemodialysis machine
- Group B（traditional hemodialysis+wearable filtrating artificial Kidney） (Experimental): Group B was isolated ultrafiltration with traditional dialysis machine first, and then with wearable filtrating artificial Kidney Device.
  Interventions: Device: the wearable filtrating artificial Kidney Device; Device: traditional hemodialysis machine

INTERVENTIONS:
Device: the wearable filtrating artificial Kidney Device — the wearable filtrating artificial kidney device rapidly for rapid relief of fluid overload in patients
Device: traditional hemodialysis machine — the hemodialysis machine currently used in clinical practice to reduce fluid overload in patients

SUMMARY:
Fluid overload is a common feature of diseases such as heart failure and kidney injury, which can lead to pulmonary edema or even death if not treated in time. In order to rapidly relieve fluid overload in patients, a wearable filtrating artificial kidney device was developed. The purpose of this study is to evaluation of the precision, security, and operability of wearable filtrating artificial kidney device for on-site medical rescue.

DETAILED DESCRIPTION:
Background:Fluid overload into the tissue spaces of the body can lead to damage to multiple organs, mainly the heart, kidneys, lungs, and gastrointestinal system. Fluid overload can diminish myocardial function, induce maladaptive myocardial remodeling, and decrease coronary vascular reactivity, increasing the risk of myocardial ischemia. Increased interstitial fluid decreases renal capillary blood flow, leading to renal ischemia and acute renal failure. In the lungs, excess extravascular water impairs gas exchange, decreases pulmonary compliance, and significantly increases morbidity and mortality. Fluid overload can also lead to impaired liver function and prolonged wound healing, as well as being a risk factor for intra-abdominal hypertension, and edema of the intestinal wall can lead to decreased absorption, intestinal distention, and even intestinal obstruction.A wearable filtrating artificial kidney device has been developed to address volume overload in patients, and it has been evaluated for biosafety and animal testing, and third-party testing has been completed for device performance as required by Q/WLS 10101-2020. This study proposes to conduct human trials to evaluate its performance.

Methods: This is a prospective controlled study involving patients with fluid overload requiring ultrafiltration therapy. Inclusion criteria: 1. 18 years ≤ age ≤ 70 years, regardless of gender; 2. Patients with fluid overload requiring ultrafiltration therapy; 3. Patients voluntarily participated and obtained written informed consent signed by the patient or authorized delegate. Exclusion criteria: 1. Mechanical failure of the ultrafiltration access; 2. Presence of active infection; 3. Known HIV positivity; 4. Poor compliance with the regimen; 5. Other serious diseases, such as active or previously treated residual malignancy or systemic infection, cirrhosis, anemia (Hb < 70 g/L), and intractable hypertension. 6. History of alcohol and drug abuse (meaning use of illicit drugs); 7. Women of childbearing age who are pregnant or breastfeeding and do not agree to use effective contraception during the trial; 8. Any other condition that, in the opinion of the investigator, prevents the patient from participating in the trial.Primary Outcome Measure:(1)Precision of ultrafiltration:Ultrafiltration volume precision, ultrafiltration speed precision;(2).Security:Pressure alarm (times), bubble monitoring (times), sound and light alarm (times) and other machine indicators;patients' complaints of improvement, tolerance, comfort, etc.(3).Operability:Human-machine interaction, friendly interface, battery life, overall mass, main volume, portable features, etc.SPSS is applied for statistical analysis, and continuous variables are expressed as mean±standard deviation, and non-continuous variables are expressed as percentages. Comparisons between the two data are made by independent t-test or χ2 test, and P<0.05 is statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1.18 years ≤ age ≤ 70 years, regardless of gender. 2.Patients with fluid overload requiring ultrafiltration therapy. 3.The patient voluntarily participates and has obtained written informed consent signed by the patient or authorized delegate.

Exclusion Criteria:

1. Mechanical failure of the ultrafiltration access.
2. Presence of an active infection.
3. Known HIV positivity.
4. Poor compliance and inability to follow the regimen.
5. Other serious medical conditions such as active, or previously treated residual malignancy or systemic infection, cirrhosis, anemia (Hb<70g/L), intractable hypertension, etc.
6. History of alcohol and drug abuse (defined as the use of illegal drugs)
7. Pregnancy or breastfeeding, women of childbearing age who do not agree to use effective contraception for the duration of the trial
8. Any other condition that, in the opinion of the investigator, prevents the patient from enrolling in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-06-25 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ultrafiltration volume of device | 4 hours
  Compare the ultrafiltration volume of wearable filtrating artificial Kidney and traditional hemodialysis machine
ultrafiltration speed of device | 4 hours
  Compare the ultrafiltration speed of wearable filtrating artificial Kidney and traditional hemodialysis machine

SECONDARY OUTCOMES:
incidence of alarms of device | 4 hours
  Compare the incidence of alarms of wearable filtrating artificial Kidney and traditional hemodialysis machine
arterial pressure displayed by the device | 4 hours
  Compare the arterial pressure displayed by wearable filtrating artificial Kidney and traditional hemodialysis machine
venous pressure displayed by the device | 4 hours
  Compare the venous pressure displayed by wearable filtrating artificial Kidney and traditional hemodialysis machine
patient satisfaction with the device | 4 hours
  Survey question asking for qualitative description of satisfaction
nurse satisfaction with the device | 4 hours
  Survey question asking for qualitative description of satisfaction
weight of device | before hemodialysis
  The weight of device is measured in kg
volume of device | before hemodialysis
  The volume of device is measured in Length x width x height

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China